CLINICAL TRIAL: NCT06442280
Title: Enhanced Diuresis and Natriuresis in Acute Decompensated Heart Failure Patients Treated With SGLT-2 Inhibitor and High-Dose Furosemide Plus Small-Volume Hypertonic Saline Solution: A Clinical Trial
Brief Title: SGLT-2 Inhibitor and High-Dose Furosemide Plus Small-Volume Hypertonic Saline Solution in Acute HF
Acronym: DAPA-TONIC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPalermo7
Record Dates: First submitted 2024-01-19; First posted 2024-06-04 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure Acute; Diabetes Type 2; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction
Keywords: Acute Heart Failure; Diabetes Type 2; SGLT-2 inhibitors; Furosemide; Hypertonic Solution
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Saline Solution, Hypertonic; Furosemide

STUDY DESIGN:
Intervention Model Description: Patients will be categorized into 4 groups: the first group will undergo 15 minutes intravenous infusion of furosemide combined with hypertonic saline solution (100 mL) twice daily along with severe water restriction (< 500 mL); the second group will receive intravenous furosemide as a bolus twice daily and severe water restriction (< 500 mL) without hypertonic saline solution; the third group will undergo 15 minutes intravenous infusion of furosemide combined with hypertonic saline solution (100 mL) twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin); the fourth group will receive intravenous furosemide as a bolus without hypertonic saline solution twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dapa-Tonic (Experimental): This group will undergo a 15-minute intravenous infusion of furosemide combined with hypertonic saline solutions (100 mL) twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin).
  Interventions: Drug: Dapagliflozin tablet; Drug: Hypertonic Saline Solution, 1 Ml
- Tonic-Placebo (Placebo Comparator): This group will undergo a 15-minute intravenous infusion of furosemide combined with hypertonic saline solutions (100 mL) twice daily along with severe water restriction (< 500 mL).
  Interventions: Drug: Hypertonic Saline Solution, 1 Ml
- Furosemide-Placebo (Placebo Comparator): This group will undergo intravenous furosemide twice daily and severe water restriction (< 500 mL) without hypertonic saline solutions.
  Interventions: Drug: Furosemide Injection
- Dapa-Furo (Active Comparator): This group will undergo intravenous furosemide without hypertonic saline solutions twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin).
  Interventions: Drug: Dapagliflozin tablet; Drug: Furosemide Injection

INTERVENTIONS:
Drug: Dapagliflozin tablet — Dapagliflozin 10 mg 1 tablet once daily
  Other Names: SGLT2 inhibitor
  Arms: Dapa-Furo; Dapa-Tonic
Drug: Hypertonic Saline Solution, 1 Ml — Intravenous infusion of furosemide combined with hypertonic saline solutions (100 mL) twice daily
  Other Names: Hypertonic Solution, Saline
  Arms: Dapa-Tonic; Tonic-Placebo
Drug: Furosemide Injection — Furosemide 20 mg
  Other Names: FUROSEMIDE
  Arms: Dapa-Furo; Furosemide-Placebo

SUMMARY:
The purpose of the current investigation is to demonstrate the efficacy of high-dose furosemide plus small-volume hypertonic saline solution and a Sodium-Glucose cotransporter-2 (SGLT-2) inhibitor among patients admitted for acute exacerbation of heart failure, in determining a significant increase in diuresis and natriuresis. It is also accompanied by a rapid reduction in body weight and a substantial decrease in hospitalization length without compromising renal function.

DETAILED DESCRIPTION:
All enrolled patients will undergo a comprehensive physical examination post-randomization. This examination will involve a meticulous assessment of congestive heart failure (CHF) indicators, encompassing the measurement of bodyweight (BW) (taken in the morning before breakfast), supine and standing blood pressure (BP [average of 3 readings]), and heart rate (HR). Fasting blood samples will be collected daily throughout the hospital stay to ascertain serum laboratory parameters (creatinine, sodium, potassium, and N-terminal pro b-type natriuretic peptide) until achieving a clinically stabilized condition. Urine output will be measured daily, also to detect creatinine, sodium, potassium urinary levels and glycosuria. Additionally, an electrocardiogram and echocardiogram (to derive EF using the modified Simpson rule with 2 cross-sectional views [4- and 2-chamber apical views], right atrium volume (RA volume, ml/m2), left atrial volume (LA volume ml/m2), inferior vena cava diameter (IVC diameter, cm), interventricular septum thickness at end-diastole (IVSd, cm), right ventricular basal diameter at end-diastole (RVD1 basal, mm), right ventricular mid diameter at end-diastole (RVD2 mid, mm), right ventricular longitudinal diameter at end-diastole (RVD3 long, mm), right ventricular outflow tract at proximal and distal (RVOT prox and distal, mm), fractional area change (FAC, %), E wave dominant (m/s), A wave dominant (m/s), tricuspid valve E/A wave ratio (E/ATrV), tissue Doppler echocardiography (TDE, ms), eak velocity in early diastole of tricuspid annulus (TDI) (m/s), tricuspid valve e'/a' ratio (TDI, m/s), peak systolic velocity tricuspid annulus (Pulsed TDI, m/s) will be conducted prior to hospital discharge.

Patients will be categorized into 4 groups: the first group will undergo 15 minutes intravenous infusion of furosemide combined with hypertonic saline solutions (100 mL) twice daily along with severe water restriction (< 500 mL); the second group will receive intravenous furosemide as a bolus twice daily and severe water restriction (< 500 mL) without hypertonic saline solutions; the third group will undergo 15 minutes intravenous infusion of furosemide combined with hypertonic saline solutions (100 mL) twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin); the fourth group will receive intravenous furosemide as a bolus without hypertonic saline solutions twice daily, severe water restriction (< 500 mL), and SGLT2 inhibitors (Dapagliflozin). The groups will maintain a normal sodium intake (120 mmol/day). The daily furosemide dosage will be determined based on diuretic requirements, urinary output, BP readings, and the severity of congestion signs and symptoms. The hypertonic saline solutions dosage for each patient (in groups 1 and 3) will be determined following these guidelines: for serum Na values of 125 milliequivalent/L, the hypertonic saline solutions concentration will be 4.6%; for serum Na values between 126 and 135 milliequivalent/L, the hypertonic saline solutions concentration will be 3.5%; and for serum Na values of 135 milliequivalent/L, the hypertonic saline solutions concentration will range between 1.4% and 2.4%. Throughout the study period, patients diagnosed with Heart Failure with Reduced Ejection Fraction (HFrEF) will receive angiotensin converting enzyme inhibitors, sartans, angiotensin receptor-neprilysin inhibitors, beta blockers, and mineralocorticoid inhibitors. The objective is to optimize heart failure therapy in alignment with the most recent European Society of Cardiology guidelines published in August 2023. Daily, there will be meticulous monitoring of body weight (in the morning before breakfast) and 24-hour urinary volume measurements. Serum and urinary laboratory parameters will be assessed daily until achieving a clinically stabilized condition, defined as a shift in New York Heart Association functional class to at least second b and reaching the ideal body weight calculated via the Lorenz formula. Upon attaining this clinically stabilized state, intravenous administration of furosemide and hypertonic saline solutions will cease, transitioning to oral furosemide administration, while maintaining the unchanged optimal therapy post-discharge according to the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* acute heart failure;
* diabetes type 2.

Exclusion Criteria:

* low estimated glomerular filtration rate;
* hypernatremia;
* diabetes type 1;
* non-cardiac causes of dyspnea;
* cardiogenic shock;
* recent occurrence of Acute Coronary Syndrome;
* ketoacidosis;
* hyperosmolar hyperglycemic syndrome.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Diuresis from the baseline and up to 1 week | an average of 1 week
  Daily urinary volume (mL) are detected by chemiluminescence immunoassay.
Natriuresis from the baseline and up to 1 week | an average of 1 week
  Daily natriuresis (mEq/L) are detected by chemiluminescence immunoassay.
Length of hospital stay | immediately after the intervention
  Duration of hospital stay in days.

SECONDARY OUTCOMES:
Kidney function during treatment | an average of 1 week
  Daily evaluation of creatinine (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Miceli, PhD, Principal Investigator — A.O.U.P. Paolo Giaccone Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Liszkowski M, Nohria A. Rubbing salt into wounds: hypertonic saline to assist with volume removal in heart failure. Curr Heart Fail Rep. 2010 Sep;7(3):134-9. doi: 10.1007/s11897-010-0018-4. PMID 20607462
- [Result] Arrigo M, Jessup M, Mullens W, Reza N, Shah AM, Sliwa K, Mebazaa A. Acute heart failure. Nat Rev Dis Primers. 2020 Mar 5;6(1):16. doi: 10.1038/s41572-020-0151-7. PMID 32139695
- [Result] Parrinello G, Di Pasquale P, Torres D, Cardillo M, Schimmenti C, Lupo U, Iatrino R, Petrantoni R, Montaina C, Giambanco S, Paterna S. Troponin I release after intravenous treatment with high furosemide doses plus hypertonic saline solution in decompensated heart failure trial (Tra-HSS-Fur). Am Heart J. 2012 Sep;164(3):351-7. doi: 10.1016/j.ahj.2012.05.025. Epub 2012 Aug 17. PMID 22980301
- [Result] Parrinello G, Paterna S, Di Pasquale P, Torres D, Mezzero M, Cardillo M, Fasullo S, La Rocca G, Licata G. Changes in estimating echocardiography pulmonary capillary wedge pressure after hypersaline plus furosemide versus furosemide alone in decompensated heart failure. J Card Fail. 2011 Apr;17(4):331-9. doi: 10.1016/j.cardfail.2010.11.003. Epub 2010 Dec 24. PMID 21440872
- [Result] Paterna S, Di Pasquale P, Parrinello G, Fornaciari E, Di Gaudio F, Fasullo S, Giammanco M, Sarullo FM, Licata G. Changes in brain natriuretic peptide levels and bioelectrical impedance measurements after treatment with high-dose furosemide and hypertonic saline solution versus high-dose furosemide alone in refractory congestive heart failure: a double-blind study. J Am Coll Cardiol. 2005 Jun 21;45(12):1997-2003. doi: 10.1016/j.jacc.2005.01.059. PMID 15963399
- [Result] Xie Y, Wei Y, Li D, Pu J, Ding H, Zhang X. Mechanisms of SGLT2 Inhibitors in Heart Failure and Their Clinical Value. J Cardiovasc Pharmacol. 2023 Jan 1;81(1):4-14. doi: 10.1097/FJC.0000000000001380. PMID 36607775
- [Result] Solomon SD, Vaduganathan M, Claggett BL, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Belohlavek J, Chiang CE, Willem Borleffs CJ, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Kerr Saraiva JF, Tereschenko SN, Thierer J, Vardeny O, Verma S, Vinh PN, Wilderang U, Zaozerska N, Lindholm D, Petersson M, McMurray JJV. Baseline Characteristics of Patients With HF With Mildly Reduced and Preserved Ejection Fraction: DELIVER Trial. JACC Heart Fail. 2022 Mar;10(3):184-197. doi: 10.1016/j.jchf.2021.11.006. PMID 35241246
- [Result] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Result] Ostermann M, Bellomo R, Burdmann EA, Doi K, Endre ZH, Goldstein SL, Kane-Gill SL, Liu KD, Prowle JR, Shaw AD, Srisawat N, Cheung M, Jadoul M, Winkelmayer WC, Kellum JA; Conference Participants. Controversies in acute kidney injury: conclusions from a Kidney Disease: Improving Global Outcomes (KDIGO) Conference. Kidney Int. 2020 Aug;98(2):294-309. doi: 10.1016/j.kint.2020.04.020. Epub 2020 Apr 26. PMID 32709292
- [Result] Clark WF, Sontrop JM, Macnab JJ, Suri RS, Moist L, Salvadori M, Garg AX. Urine volume and change in estimated GFR in a community-based cohort study. Clin J Am Soc Nephrol. 2011 Nov;6(11):2634-41. doi: 10.2215/CJN.01990211. Epub 2011 Sep 1. PMID 21885793
- [Result] Oh SW, Han SY. Loop Diuretics in Clinical Practice. Electrolyte Blood Press. 2015 Jun;13(1):17-21. doi: 10.5049/EBP.2015.13.1.17. Epub 2015 Jun 30. PMID 26240596